CLINICAL TRIAL: NCT03299231
Title: Oscillating Positive Expiratory Pressure Device for Mucous Clearing in Severe Exacerbation of COPD Requiring Hospitalization Targeting Outcome: A Randomized, Double Blind, Sham Controlled Trial (SIMPLE)
Brief Title: Oscillating Positive Expiratory Pressure Devices and Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: SIMPLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Trudell Medical International (Industry)
Responsible Party: Principal Investigator, Hesham Raafat, Ass. Professor of chest medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU P56/2017
Record Dates: First submitted 2017-09-22; First posted 2017-10-03 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; acute exacerbation; OPEP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, Parallel group (1:1), Randomized, double blind, sham controlled, single center.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization carried by a third party not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobika (Active Comparator): Group of participants with COPD, hospitalized for severe exacerbation and using the active oscillating positive expiratory pressure device (OPEP). The device is a hand held one. Used mostly in subjects with bronchiectasis for mucus clearing. Estimated number of subjects in this arm is 80. The device has an adjustable resistance which will be set by a health care provider in the study team. The device is to be used three times daily from 10 to 20 minutes according to subject's effort.
  Interventions: Device: OPEP Aerobika
- Sham device (Sham Comparator): Group of participants using the same looking device which is devoid from nebulizer port valve so it is not functioning (sham device). The sham arm is a control arm. It will be used as the active comparator three times daily for 10 to 20 minutes according to subject's effort
  Interventions: Device: OPEP Aerobika Sham device

INTERVENTIONS:
Device: OPEP Aerobika — Previous studies of OPEP device shows preliminary benefit in subjects with COPD. No serious adverse events were recorded in previous studies. The device is FDA registered.
  Arms: Aerobika
Device: OPEP Aerobika Sham device — The same OPEP device which is devoid of the nebulizer port valve to render it inactive. Used for control sham arm.
  Arms: Sham device

SUMMARY:
Sputum production increases in acute exacerbation of COPD, both in amount and consistency. It increases airways obstruction and hence delays improvement and prolongs hospital stay. oscillating positive expiratory pressure (OPEP) devices were extensively studied in cystic fibrosis and bronchiectasis. Only seldom studied in chronic bronchitis. This study aims to measure the effects of mucous clearing device in hospitalized patients with acute exacerbation of COPD.

DETAILED DESCRIPTION:
In this study, investigators will investigate the change of objective measurements of lung functions and exercise capacity in addition to subjective measures of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients, stages 3-4 according to GOLD guidelines 2016, with post bronchodilator FEV1/FVC < 70% of predicted and FEV1 < 50% with exacerbations necessitates hospital admission.
* Smokers or Ex-smokers.
* Able and willing to provide informed signed consent. Able and understanding the correct use of the bronchial clearing device.
* Able to perform effectively spirometry.
* Able and willing to receive the management plane as indicated including systemic steroids if seemed necessary.

Exclusion Criteria:

* Other obstructive pulmonary diseases or those do not fulfill the criteria of COPD diagnosis.
* Nonsmokers.
* Presence of major comorbidity causing organ dysfunction as cardiac (including severe pulmonary hypertension), renal, or liver impairment (not including diabetes, arterial hypertension, or obesity).
* Presence of lobar pneumonia.
* Suspicion of bronchogenic malignancy.
* Any other complication either at admission or during hospital stay as pneumothorax, pulmonary embolism, myocardial infarction, acute coronary syndrome, cerebrovascular accidents, ...
* Patients unable or not willing to provide informed signed consent.
* Patients unable to use the bronchial clearing device.
* Patients unable to perform spirometry.
* Patients unable or not willing to comply to the management plan or the study protocol.
* Patients receiving regular oral steroids or non-selective beta blockers.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
percent change of Forced expiratory volume in first second (FEV1) | at 12 weeks after hospital discharge
  change in volume of air expired forcefully in first second of expiration
percent change of Forced vital capacity (FVC) | at 12 weeks after hospital discharge
  change in total volume of air expired forcefully
percent change of six minutes walking distance (6MWD) | at 12 weeks after hospital discharge
  distance in meters a subject walk within 6 minutes

SECONDARY OUTCOMES:
change in health related quality of life | 12 weeks after hospital discharge
  measured by Saint George Respiratory Questionnaire
change in score of shortness of breath | 12 weeks after hospital discharge
  measure by baseline and transitional dyspnea index
hospital stay | first day of hospital admission to day of hospital discharge up to 12 weeks
  measured in days of hospital stay
hospital readmission | 4 weeks after discharge
  admission to hospital after 30 days of discharge due to COPD exacerbation
severe COPD exacerbation | 12 weeks after discharge
  exacerbation of COPD need hospitalization
Moderate COPD exacerbation | 12 weeks after discharge
  exacerbation of COPD need additional treatment as antibiotics and/or steroids

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kushnarev, Study Director — Trudell Medical International; Hesham H Raafat, M.D., Principal Investigator — Ain Shams University; Yasser Mostafa, M.D., Study Director — Ain Shams University; Brian W Carlin, Study Director — West Penn Allegheny Health System
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No